CLINICAL TRIAL: NCT03967691
Title: IL-6 Regulation of Substrate Metabolism and Influence of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Helga Ellingsgaard, Group leader, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: TOSS
Record Dates: First submitted 2019-05-22; First posted 2019-05-30 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Obesity; Healthy
Keywords: Interleukin-6; Tocilizumab; Exercise; Substrate Metabolism; Lipolysis
MeSH Terms: conditions — Obesity; Motor Activity | interventions — tocilizumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study is designed in a placebo-controlled crossover manner, consisting of a screening visit and three study visits/study days. the Subjects will be infused with saline (placebo) on two of the study days and tocilizumab on one of the study days.
Who Masked: Participant
Masking Description: Only subjects will be masked regarding order of saline and tocilizumab infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Saline infusion (Placebo Comparator): Subjects will be infused with saline (placebo) on study day 1
  Interventions: Drug: Saline 0.9%
- Tocilizumab infusion (Active Comparator): Subjects will be infused with tocilizumab on study day 2
  Interventions: Drug: Tocilizumab infusion
- Saline infusion under tocilizumab influence (Other): Subjects will be infused withsaline (but still under the influence of tocilizumab) on study day 3
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Tocilizumab infusion — Tocilizumab (8mg/kg body weight diluted to 100 ml NaCl 0.9%) will be infused over 1 hour
  Other Names: RoActemra
  Arms: Tocilizumab infusion
Drug: Saline 0.9% — 100 ml NaCl 0.9% will be infused over 1 hour
  Other Names: Saline
  Arms: Saline infusion; Saline infusion under tocilizumab influence

SUMMARY:
The aim of the study is to investigate the effects of blocking IL-6 signaling with tocilizumab on lipid, glucose and protein metabolism during rest and exercise in healthy and obese humans.

Interleukin-6 is a molecule produced by a variety of cells and impacts on energy metabolism during fasting and fed conditions. Systemic IL-6 levels are low but increase acutely in response to fasting, exercise and infection, and also chronically in response to obesity and other conditions of lowgrade inflammation.Our recent human intervention study showed that IL-6 receptor blockade prevents exercise training from reducing visceral fat mass.

Whether IL-6 receptor blockade directly regulates lipolysis and/or lipid oxidation in humans is however unclear. Therefore, this study will be performed to investigate the physiological role of IL-6 on lipid, glucose and protein metabolism in humans.

DETAILED DESCRIPTION:
The aim of the study is to assess changes in substrate kinetics, that is, lipolytic rate, rate of appearance and disappearance of free fatty acids, fatty acid oxidation, glucose rate of appearance and disappearance and protein synthesis and degradation during rest and exercise with and without IL-6 receptor blockade. We will assess the acute effects of blocking IL-6 as well as the long-term consequences of IL-6 receptor blockade on all the above parameters.

Overall, we hypothesize that blocking IL-6 changes substrate kinetics. More specifically we hypothesize that blocking IL-6 reduces the appearance of free fatty acids, reduces the lipolytic rate and lipid oxidation. We hypothesize that the consequences of blocking IL-6 will be observed during resting and exercising conditions and both immediately and longterm after IL-6 receptor blockade. We hypothesize that IL-6 receptor blockade results in an increased respiratory exchange ratio (RER) and thus increased reliance on glucose as substrate.

In this study 10 healthy males and 10 obese males will be included. Subjects will be infused with saline on 2 of the study days and tocilizumab on 1 of the study days.

Isotope dilution techniques with [6,6-2H2]Glucose, [1,1,2,3,3-D5]glycerol, K-[U-13C16]palmitate, L-[ring-D5]phenylalanine, L-[D2]tyrosine will be applied to assess lipid, glucose and protein kinetics. Respiratory exchange ratio will be measured by indirect calorimetry. The BORG scale will be used to assess the perceived exertion during exercise.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 18 and > 25 kg/m2 or ≥ 30 and ≤ 40 kg/m2
* Healthy (based on screening)

Exclusion Criteria:

* Smoking
* Severe thyroid or heart disease
* inflammatory diseases
* current infection
* liver disease
* kidney disease
* immunosuppressive disease
* corticosteroid use
* regular NSAID usage
* aspirin use >100 mg/d
* history of carcinoma
* history of tuberculosis
* anemia
* neutropenia
* low platelets
* bleeding disorders
* obstructive pulmonary disease

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Lipolytic rate | 0-28 days
  Rate of appearance and disappearance of glycerol and palmitate, fatty acid oxidation during rest and exercise in the presence of tocilizumab as compared to placebo

SECONDARY OUTCOMES:
Glucose kinetics | 0-28 days
  Rate of appearance and disappearance of glucose during rest and exercise in the presence of tocilizumab as compared to placebo
Protein metabolism | 0-28 days
  Rate of appearance and disappearance of phenylalanine and tyrosine during rest and exercise in the presence of tocilizumab as compared to placebo
Respiratory exchange ratio (RER) | 0-28 days
  RER during rest and exercise in the presence of tocilizumab as compared to placebo
Perceived exhaustion during exercise | 0-28 days
  Borg scale (rate of perceived exertion during exercise; score range from minimum 6 to maximum 20; 6 = "no feeling of exertion", 20 = "very, very hard") in the presence of tocilizumab as compared to placebo
Glucose | 0-28 days
  Change in glucose during rest and exercise in the presence of tocilizumab as compared to placebo
Insulin | 0-28 days
  Changes in insulin during rest and exercise in the presence of tocilizumab as compared to placebo
C-peptide | 0-28 days
  Change in c-peptide during rest and exercise in the presence of tocilizumab as compared to placebo
Glucagon | 0-28 days
  Change in glucagon during rest and exercise in the presence of tocilizumab as compared to placebo
Cortisol | 0-28 days
  Change in cortisol during rest and exercise in the presence of tocilizumab as compared to placebo
Adrenaline | 0-28 days
  Change in adrenaline during rest and exercise in the presence of tocilizumab as compared to placebo
Noradrenaline | 0-28 days
  Changes in noradrenaline during rest and exercise in the presence of tocilizumab as compared to placebo
Interleukin 6 | 0-28 days
  Change in IL-6 during rest and exercise in the presence of tocilizumab as compared to placebo
Free fatty acids | 0-28 days
  Change in free fatty acids during rest and exercise in the presence of tocilizumab as compared to placebo
Triglycerides | 0-28 days
  Changes in triglycerides during rest and exercise in the presence of tocilizumab as compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Helga Ellingsgaard, Ph.D., Principal Investigator — CFAS, Rigshospitalet
Locations (1):
- Rigshospitalet, Centre of Inflammation and Metabolism (CIM) Centre for Physical Activity Research (CFAS), Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trinh B, Peletier M, Simonsen C, Plomgaard P, Karstoft K, Pedersen BK, van Hall G, Ellingsgaard H. Amino Acid Metabolism and Protein Turnover in Lean and Obese Humans During Exercise-Effect of IL-6 Receptor Blockade. J Clin Endocrinol Metab. 2022 Jun 16;107(7):1854-1864. doi: 10.1210/clinem/dgac239. PMID 35442403
- [Derived] Trinh B, Peletier M, Simonsen C, Plomgaard P, Karstoft K, Klarlund Pedersen B, van Hall G, Ellingsgaard H. Blocking endogenous IL-6 impairs mobilization of free fatty acids during rest and exercise in lean and obese men. Cell Rep Med. 2021 Sep 9;2(9):100396. doi: 10.1016/j.xcrm.2021.100396. eCollection 2021 Sep 21. PMID 34622233